CLINICAL TRIAL: NCT06802991
Title: Optimised Post-discharge Care in Older Patients After Surgery for Colon Cancer (ERAS 3.0)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Elna A. Dalsgaard, MSc, ph.d. student, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-24078496
Record Dates: First submitted 2025-01-19; First posted 2025-01-31 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-01

CONDITIONS: Colon Cancer; Frailty
Keywords: ERAS 3.0; colon cancer surgery; comprehensive geriatric assessment
MeSH Terms: conditions — Colonic Neoplasms; Frailty | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS 3.0 group (Experimental): Post-surgery support at discharge and at home
  Interventions: Other: ERAS 3.0 (Enhanced Recovery After Surgery)
- Standard care group (No Intervention): Standard care, which is no support after discharge

INTERVENTIONS:
Other: ERAS 3.0 (Enhanced Recovery After Surgery) — Nutritional support at discharge and home visits which include comprehensive geriatric assessment, nutritional guidance by dietitian, and instructions on exercise and physical activity.
  Arms: ERAS 3.0 group

SUMMARY:
The purpose of the study is to investigate whether an extended program (ERAS 3.0) initiated hospital discharge, can improve recovery in elderly, frail patients who have undergone surgery for colon cancer.

The study is a randomised controlled trial with two groups: an intervention group receiving the ERAS 3.0 program and a control group recieving standard care. The ERAS 3.0 program includes a comprehensive geriatric health assessment, dietary counseling from a dietitian, and instructions on training and physical activity. These activities will take place in the participant's homes after hospital discharge. Data will be collected at multiple time points: at the hospital, 12 days post-discharge (at the outpatient clinic), and at 1 and 3 months post discharge in the participants' homes.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* Clinical Frailty Scale preoperative score 4-7
* Nutritional Risk Screening tool (NRS 2002) > 3
* Elective colonic resection
* No stoma planned
* Minimally invasive surgical approach (laparoscopic or robotic)
* Patients discharged to own home
* Informed consent to participate

Exclusion Criteria:

* Stoma creation during index surgery
* Conversion to laparotomy
* Major complications following surgery (Clavien-Dindo >3a)
* Participation in other randomised trials in conflict with the protocol and end- points of the ERAS 3.0 project
* Discharged with tube feeding and parenteral nutrition (partially or completely)
* Known food allergies to dairy or any other ingredient contained in the nutrition package
* Incapable of providing informed consent
* Discharge to 24-hour municipal rehabilitation facility
* All conditions including psychological, geographical, and social factors that could hinder adherence to the trial protocol
* Neoadjuvant radio- or chemotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative recovery | 10-14 days after surgery
  Postoperative recovery is measured as a change in the Quality of Recovery-15 questionnaire. Through 15 questions, the time spent in common postoperative conditions during the last 24 hours is estimated. Each question has a scale from 0 to 10, resulting in a maximum total score of 150.

SECONDARY OUTCOMES:
Health realted Quality of Life (HrQoL) | 12, 30 and 90 days after surgery
  HrQoL will be measured using the EQ-5D-5L questionnaire. The EQ-5D-5L questionnaire comprises five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain has five response categories, ranging from having no problems to being unable to perform the activity. The responses are converted into a utility index value, reflecting health status compared to the reference of the general population (norm data). A visual analogue scale (VAS) is also included, where health is rated on a scale from 0 (worst health you can imagine) to 100 (best health you can imagine). Permission will be sought to use the tool.
Postoperative recovery | 30 and 90 days after surgery
  Postoperative recovery is measured as a change in the Quality of Recovery-15 questionnaire. Through 15 questions, the time spent in common postoperative conditions during the last 24 hours is estimated. Each question has a scale from 0 to 10, resulting in a maximum total score of 150.
Activities of daily living | 12, 30 and 90 days after surgery
  Activities in daily living are assessed using the Functional Recovery Score (FRS) to evaluate functional recovery after surgery. The eleven-item questionnaire comprises three main components: basic activities of daily living (BADL), assessed by four items; instrumental activities of daily living (IADL), assessed by six items; and mobility, assessed by one item. BADL accounts for 44 percent of the score, IADL for 23 percent, and mobility for 33 percent. Complete independence results in a score of 100 percent.
Energy- and protein intake | 12, 30 and 90 days after surgery
  Energy and protein intake will be estimated using the 24-hour dietary recall interview method. The interviews will be conducted by the investigator working on the study. The foods and drinks will be entered into the software program Vitakost to calculate the intake of protein (g) and energy (kJ) and liquid (mL). The participant's body weight will be used to calculate the intake per kilogram of body weight. The cut-off for suspecting underreporting will be evaluated retrospectively on an individual basis, taking into account any illness, readmissions, loss of body weight, activity level etc.
Appetite | 12, 30 and 90 days after surgery
  Appetite will be assessed using the Simplified Nutritional Appetite Questionnaire (SNAQ), which consists of four questions adressing appetite, taste, satiety, and meal frequency. Each question offers five possible answers, and participants select the category that best reflects their current situation. The total score ranges from 5 to 20.
Weight | 12, 30 and 90 days after surgery
Physical function and muscle strenght | 12, 30 and 90 days after surgery
  Physical function and muscle strength will be assessed using the 30-second chair stand test (30s CST), which measures the number of times an individual can rise from and sit down in a standardized chair within 30 seconds. To accommodate participants' abilities, the chair stand test will be modified according to three versions as needed.
Muscle mass by BIA | 12, 30 and 90 days after surgery as well as 1 (CT) and 3 (CT) years after surgery
  Total and appendicular muscle mass (kg and percent) will be measured by bioelectrical impedance analysis (BIA). This method involves passing a low-level electrical current through the body to measure electrical impedance, or resistance, encountered by the current as it flows through different tissues. Tissues rich in electrolyte-containing water, such as skeletal muscle, have lower resistance and thus higher conductivity. Conductivity is directly proportional to total body water. Lean muscle mass is derived from the conductivity measurement, and fat mass (in kilograms and percentage) is subsequently calculated by subtracting lean muscle mass from total body weight.
  Body weight and height are entered manually to aid in calculations.
Rate of readmission | within 30 days after discharge
  Readmission rate is defined as any unplanned hospitalisation within 30 days after discharge from hospital.
Postoperative complications | within 30 and 90 days after discharge
  The occurrence of post-operative complications, including infections requiring treatment within 30 and 90 days will be registered numerically.
Number of reoperations | within 1 and 6 months after discharge
  The occurence of reoperations will be registered
Total length of hospital stay | within 6 months after discharge
Days alive and out of the hospital | within 30 and 90 days after discharge
Mortality | Within 1, 3, 6, and 12 months after primary surgery
Muscle mass by CT | at baseline, after one and three years
  Muscle mass by will be measured by computed tomography (CT) scan. All CT scans are part of routine care concerning the cancer disease and are therefore not research-related add-ons to routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Professor, dr. med., Study Director — Center of Perioperative Optimisation, Copenhagen University Hospital at Herlev
Locations (1):
- University Hospital Herlev, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munk T, Svendsen JA, Knudsen AW, Ostergaard TB, Thomsen T, Olesen SS, Rasmussen HH, Beck AM. A multimodal nutritional intervention after discharge improves quality of life and physical function in older patients - a randomized controlled trial. Clin Nutr. 2021 Nov;40(11):5500-5510. doi: 10.1016/j.clnu.2021.09.029. Epub 2021 Sep 24. PMID 34656032
- [Background] Dolin TG, Mikkelsen M, Jakobsen HL, Nordentoft T, Pedersen TS, Vinther A, Zerahn B, Vistisen KK, Suetta C, Nielsen D, Johansen JS, Lund CM. Geriatric assessment and intervention in older vulnerable patients undergoing surgery for colorectal cancer: a protocol for a randomised controlled trial (GEPOC trial). BMC Geriatr. 2021 Jan 30;21(1):88. doi: 10.1186/s12877-021-02045-9. PMID 33516195